CLINICAL TRIAL: NCT06441123
Title: Development of a New Family of HIV Latency Regulators (LRAs) Targeting the Tat Viral Protein
Acronym: TatLat
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0276
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
Keywords: HIV-1; Tat; latency; latency reversing agents; transcription
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 ml of blood (5 tubes of 4 ml each) from 24 people living with HIV who are on AntiRetroviral Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Blood Sampling — 20 ml of blood (5 tubes of 4 ml) will be collected once.

SUMMARY:
Antiretroviral therapy (ART) prevents HIV from multiplying. However, if people living with HIV stop taking ART, the virus quickly reappears in their blood due to the random activation of hidden infected cells. These hidden cells contain HIV that is not active and do not produce the virus. These cells are a major challenge in finding a cure for HIV.

One of the most promising ways to get rid of these hidden infected cells is by activating them with special drugs called latency-reversing agents (LRAs). This process, known as the "shock-and-kill" strategy, involves waking up the hidden virus ("shock" phase) so that it can be destroyed by the body's immune system or by the virus itself ("kill" phase).

Investigators are developing new LRAs that target and activate a viral protein called Tat, which is necessary for the virus to start producing again and for reversing its dormant state.The lead compound, named D10, is the first of its kind to target the Tat protein. This compound has been patented and has shown activity in activating the virus in lab-grown cells. Now, investigators need to test its effectiveness on real target cells from people living with HIV.

DETAILED DESCRIPTION:
20 ml of blood (5 tubes of 4 ml each) will be collected from 24 people living with HIV who are on ART. The inclusion criteria for this study are: being HIV-positive, having an undetectable viral load for more than 12 months, and having a history of very low T-CD4 counts (nadir < 200 cells/mm³).

In the lab, investigators will isolate immune cells (PBMCs) from the blood using a special technique. These cells will then be placed in small wells and treated with LRAs for 18-20 hours. Investigators will measure the virus produced in the cell supernatant using two methods: q-RT-PCR for viral RNA and p24 ELISA for viral protein. The results will be analyzed using conventional statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* HIV-positive
* On ART (antiretroviral therapy)
* HIV-1 RNA undetectable for more than 12 months
* Nadir CD4 count < 200/µL

Exclusion Criteria:

* Lack of antiretroviral treatment
* Immunosuppressive treatments
* History of cancer less than 5 years old
* Pregnant or breast-feeding women
* Persons protected by law (under guardianship or curators), persons under court protection
* Participating in another research project with an ongoing exclusion period
* Refusal to participate in research
* Subject not affiliated to a social security scheme, or not benefiting from such a scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is aviremic HIV-positive individuals, with no age criterion, having a long history of HIV infection (nadir < 200 CD4/µL
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Quantity of p24 in the cell supernatant 18-20 hours after the addition of the LRAs (Latency Reversing Agents) | INCLUSION VISIT
  Viral production is considered significant if the signal obtained from the p24 ELISA of these supernatants is more than twice the background observed in the absence of LRA

SECONDARY OUTCOMES:
Quantity of viral RNA in the cell supernatant 18-20 hours after the addition of LRAs. | INCLUSION VISIT
  quantity of viral RNA in the cell supernatant 18-20 hours after the addition of LRAs.
Measure the effective dose of D10 to reverse the latency of latent HIV-infected PBMCs | INCLUSION VISIT
  effective dose of D10 to reverse the latency of latent HIV-infected PBMCs

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de MONTPELLIER, Montpellier, France

IPD SHARING:
Plan to Share IPD: No